CLINICAL TRIAL: NCT06083038
Title: Utilizing Continuous Glucose Monitoring (CGM) to Characterize and Manage Hyperglycemia in Patients Initiating Alpelisib
Brief Title: Utilizing Continuous Glucose Monitoring to Characterize and Manage Hyperglycemia in Patients Initiating Alpelisib
Status: Active, not recruiting | Type: Observational
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CBYL719A0US16T
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Hyperglycemia; Glucose management; Alpelisib
MeSH Terms: conditions — Breast Neoplasms; Hyperglycemia | interventions — Alpelisib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Metastatic breast cancer starting alpelisib
  Interventions: Drug: Alpelisib; Device: FreeStyle Libre 2 Continuous Glucose Monitor

INTERVENTIONS:
Drug: Alpelisib — Patients will receive standard of care alpelisib
Device: FreeStyle Libre 2 Continuous Glucose Monitor — All patients will wear Abbott FreeStyle Libre 2 system to obtain CGM data (glucoses measured every minute for 14 days). CGM monitors will be placed at least 10 days prior to starting alpelisib and continue CGM for at least 3 months while taking alpelisib.

SUMMARY:
This is a prospective, descriptive, single site, observational study in subjects receiving alpelisib for treatment of metastatic breast cancer. The purpose of the study is to characterize the impact of alpelisib on glucose control in patients with breast cancer using continuous glucose monitoring to measure glucose levels throughout the day and night. Patients will follow a hyperglycemia prevention and management regimen aimed to diminish hyperglycemia known to occur in most oncology patients starting alpelisib.

All patients will wear an Abbott FreeStyle Libre 2 system to obtain continuous glucose monitor (CGM) data (glucose measured every minute for 14 days). CGM will be placed at least 10 days prior to starting alpelisib and continue for at least 3 months while taking alpelisib.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or older with a diagnosis of metastatic breast cancer that are initiating treatment with alpelisib.
2. Must be willing and able to comply with study visits and procedures.
3. Must meet standard clinical criteria for utilization of alpelisib including hormone-receptor positive/HER2 negative cancer with the presence of a PIK3CA mutation.
4. Oncologist plans to use alpelisib until progression of disease or unacceptable toxicity.
5. Patients must receive cancer care during alpelisib treatment phase with a HealthPartners oncologist and be willing to see IDC/HealthPartners Diabetes Education for diabetes management.
6. Must have a compatible smartphone, access to a compatible smartphone, or the ability to upload CGM reader from home or bring the reader in to a medical visit at least once a month for uploading, to allow for remote management of diabetes and data collection.
7. Life expectancy of at least 3 months

Exclusion Criteria:

1. Known history of serious allergy to skin-adhesive material or previous cutaneous reaction to a continuous glucose monitor.
2. Known currently uncontrolled diabetes, defined as the most recent HbA1c over 10% or history of DKA within 6 months prior to enrollment.
3. Concurrent use of high-dose vitamin C, defined as ≥ 1g of oral vitamin C daily, or intravenous Vitamin C infusions.
4. Any other concurrent severe and/or uncontrolled medical condition that, in the opinion of the investigator, would cause unacceptable safety risk, compromise compliance with the protocol, or contraindicate participation in the study. One example being known requirement for high dose steroids at the time of possible enrollment into the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled to receive standard of care alpelisib for treatment of metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to peak glucose level following the administration of alpelisib | Up to 28 days after start of alpelisib
  Time (hr., min.) from taking alpelisib to the peak of the median glucose line of the standardize AGP/CGM report from day 21-28 after start of alpelisib. (calculated as- the average time to peak glucose on 7-day AGP profile minus avg time taking alpelisib). Primary outcome is time to peak glucose for all patients on alpelisib combined

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Cancer Research Center, Saint Louis Park, Minnesota, United States